CLINICAL TRIAL: NCT01642368
Title: The Optimum Omega -3 (003) Diet Study
Brief Title: The Optimum Omega-3 (003) Diet Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Catherine Champagne, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 11026
Record Dates: First submitted 2012-07-14; First posted 2012-07-17 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Stress, Physiological
Keywords: Omega-3 fatty acids; Omega-3 to omega-6 ratio; Cognitive response; Physical performance
MeSH Terms: interventions — Fatty Acids, Omega-3; Physical Functional Performance; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regular Diet (Placebo Comparator): If you are accepted into the study, you will be randomized into one of 3 treatment arms which only differ according to the foods consumed. All groups will receive smoothies with these diets.
  Interventions: Other: The Optimum Omega-3 Fatty Acid Feeding Study
- Medium Omega-3 Group (Active Comparator): If you are accepted into the study, you will be randomized into one of 3 treatment arms which only differ according to the foods consumed. All groups will receive smoothies with these diets.
  Interventions: Other: The Optimum Omega-3 Fatty Acid Feeding Study
- High Omega-3 Group (Active Comparator): If you are accepted into the study, you will be randomized into one of 3 treatment arms which only differ according to the foods consumed. All groups will receive smoothies with these diets.
  Interventions: Other: The Optimum Omega-3 Fatty Acid Feeding Study

INTERVENTIONS:
Other: The Optimum Omega-3 Fatty Acid Feeding Study — Assess whether swapping specific food ingredients in the diet can significantly improve polyunsaturated fatty acid blood profiles and improve a person's response to cognitive measures and physical fitness.
  Other Names: Omega-3 Fatty Acids; Omega-3 to Omega-6 Ratios; Physical performance and omega-3

SUMMARY:
The goal of the Optimum Omega-3 (OO3) Diet Study is to assess whether swapping specific food ingredients in diets can significantly change omega-3 blood profiles with 10 weeks of a 7-day menu in men and women (18-40 years old). We want to look at the effect on a person's response to cognition, satiety and physical fitness. Investigators think that low omega-6 and moderate omega-3 fatty acid diets may regulate emotional response and help to return to normal after load carrying activities. We plan to test the effects of improving overall fatty acids on emotional response, satiety, and physical fitness levels by a diet with an improved omega-3 to omega-6 diet compared to a control diet.

DETAILED DESCRIPTION:
The goal of the Optimum Omega-3 (OO3) Diet Study is to assess whether swapping specific food ingredients in components of US Military Garrison diet can significantly change blood profiles of n-3 HUFAs (highly unsaturated fatty acids) from baseline with 10 weeks of a 7-day menu in men and women (18-40 years old), and its effect on a person's response to cognitive measures, satiety and physical fitness (Adjunct Studies). The Department of Defense is interested in strategies to improve body composition of n-3 HUFAs and whether such strategies help people respond better emotionally. It is felt that low omega-6 and moderate omega-3 fatty acid diets may improve the regulation of emotional responses, and may accelerate return of muscle strength and lower limb range of motion after fatiguing exercise such as walking while carrying a heavy load. We plan to test the effects of improving overall fatty acids on cognitive response, satiety, and physical fitness levels by substituting all chicken meat, eggs, beef, oil and other ingredients in 7 days of 3 meals plus snacks with like products that have low omega-6 PUFA (and/or enhanced omega-3 PUFA) in comparison with a control diet in which the ingredients have not been replaced.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Healthy and able to perform all requirements of the study without injury.
* Body Mass Index (BMI), >18 and <30 Kg/m2 (BMI is a measure of your height and weight ratio.
* No history of cardiac problems or evidence of current heart problems.
* willing to use effective method of birth control if you are capable of bearing children.
* willing to consume menus for 10 consecutive weeks.
* willing to complete all study-related activities.
* If you are taking dietary supplements, you are willing to discontinue their use during the study.
* willing to follow the alcohol consumption restrictions during the study.
* Have access to a personal microwave and refrigerator to keep foods at the proper temperature for storage and consumption.

Exclusion Criteria:

* Have a history of gall stones or any other significant metabolic, blood, lung, neurologic (nervous system), immune, liver, kidney, or urologic (urinary system) disorders.
* Have any disease or condition that seriously affects body weight and/or body composition.
* Practice a vegan or vegetarian dietary lifestyle.
* Are gluten intolerant (allergic reaction to wheat products)
* Have a history of short-term (less than a month) treatment woth steroids within six months prior to randomization into the 003 Diet Study.
* Require regular use of medications that ma interfere with the study (other than contraceptives or other medications that have been on a stable dose for 6 months prior to the study). the study staff will review all medication criteria with you.
* Have diabetes.
* Have a history or evidence of significant gastrointestinal dysfunction.
* Chronically use laxatives, The use of stool softeners is acceptable. Use of bulking agents, if required, should remain constant.
* Have abnormal blood or urine results.
* Have evidence or recurrence of cancers within the past five years if it is thought to interfere with study participation, other than some skin cancers.
* Anticipate surgery during the study period.
* Donated blood during the month prior to study entry or plan to during the study.
* Have participated in other studies using an investigational drug during the preceding 3 months.
* Have had a fluctuation in body weight >10% (or about 15 lbs) in the preceding 2 months.
* Are taking prescription or over the counter medication or supplements for desired weight loss.
* Are taking prescription or over the counter medication or supplements for desired weight loss.
* Drink more than 4 alcoholic drinks daily or 6 on one occasion more than once a month within the past 6 months.
* Currently using cocaine, amphetamines, or other illicit substances.
* Have a psychiatric disorder that would interfere with your ability to complete the study.
* Are claustrophobic.
* Have a history of post-traumatic stress disorder, anxiety or panic attack disorders, or other psychological/fear/or anxiety disorders.
* Are unwilling or unable to follow the rigors of the data collection and clinical evaluation schedule over the study period.
* Are pregnant, breast feeding or planning to become pregnant before the end of the study.
* Are unwilling to be assigned at random to any intervention group.
* Are participating in another intervention program.
* Consume seafood more than 3 times per week in a the last 6 months (specifically tuna, salmon, and other types of fatty cold fishes or seafood).
* Use NSAIDS (asprin, ibuprofen, etc.) more than 2 times per week.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in blood levels of omega-3 fatty acids | After 12 weeks of feeding
  We expect to see an increase in blood levels of omega-3 fatty acids in participants following 12 weeks of consuming a diet high in omega-3 fatty acids and a lower content of omega-6 fatty acids for a more positive ratio of omega-3 to omega-6 and related to a variety of positive health outcomes.

SECONDARY OUTCOMES:
Increased stress resilience and improved physical performance. | After 12 weeks of feeding
  We expect to see improved cognitive and emotional measures. In addition, we anticipate improved physical performance in the load carrying and power testing at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Champagne, PhD,RDN,LDN, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States